CLINICAL TRIAL: NCT05100680
Title: Study of the Effect of 12-week Dietary Supplementation With a Multicomponent Nutritional Supplement on Nails and Skin: a Randomized, Double-blind Placebo-controlled Study
Brief Title: Study of the Effect of 12-week Dietary Supplementation With a Multicomponent Nutritional Supplement on Nails and Skin
Acronym: VISTMULTIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIST - Faculty of Applied Sciences (Other)
Collaborators: Ministry of Education, Science and Sport of Republic of Slovenia (Unknown); European Regional Development Fund (Other); Slovenian Research Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: VIST F4F MULTIK 01-2019
Record Dates: First submitted 2020-08-17; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Nail Damage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomp group (Active Comparator): Food supplement - 2 capsules / day containing together: 20 mg coenzyme Q10,500 mg methyl sulfonyl methane (MSM), 100 mg L-proline, 10 mg L-cysteine (as HCl monohydrate), 2 mg thiamine , 2.4 mg riboflavin, 19 mg niacin, 8.5 mg pantothenic acid, 2.3 mg vitamin B6, 0.15 mg, biotin, 0.0125 mg vitamin B12, 80 mg vitamin C, 5.5 mg vitamin A , 22 mg vitamin E, 10 mg zinc, 0.07 mg selenium, 1.1 mg copper.
  Interventions: Other: Multicomp
- Placebo group (Placebo Comparator): Placebo - 2 capsules / day containing modified starch
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Multicomp — Daily dietary supplementation over 12 weeks with test product: food supplement - 2 capsules / day containing together: 20 mg coenzyme Q10,500 mg methyl sulfonyl methane (MSM), 100 mg L-proline, 10 mg L-cysteine (as HCl monohydrate), 2 mg thiamine , 2.4 mg riboflavin, 19 mg niacin, 8.5 mg pantothenic acid, 2.3 mg vitamin B6, 0.15 mg, biotin, 0.0125 mg vitamin B12, 80 mg vitamin C, 5.5 mg vitamin A , 22 mg vitamin E, 10 mg zinc, 0.07 mg selenium, 1.1 mg copper.
  Arms: Multicomp group
Other: Placebo — Daily dietary supplementation over 12 weeks with placebo product: dietary supplement - 2 capsules / day, containing only modified starch.
  Arms: Placebo group

SUMMARY:
A double-blind, randomized, placebo-controlled efficacy study in one period will include 34 participants divided into two groups. One group will receive a test product (n = 22; test group; multicomponent dietary supplement including MSM and several vitamins and minerals); the other group received placebo capsules (n = 12; placebo group; only modified starch). Volunteers will take two capsules / day orally continuously daily for 12 weeks to assess the effect of these substances on nail growth and condition and skin.

ELIGIBILITY:
Inclusion Criteria:

* women and men who are diagnosed at the introductory term with any of the following signs of brittle nails on at least one of the assessed nails (preferably at least two signs):

  * rough surface of the nail plate or presence of keratin granulation (trachyonychia)
  * lamellar stratification - horizontal layering / peeling (onychoschizia)
  * longitudinal stratification or splitting of the distal edge, rupture (onychorrhexis)
* generally healthy
* willingness to participate in research
* signed statement of conscious and free consent to research - informed consent
* willingness not to use any dietary supplements with the active substances contained in the test product (CoQ10, biotin, niacin, vitamin C, β-carotene, vitamin E, zinc, selenium, copper, MSM, L-cysteine, L- proline), other than those to be allocated by researchers
* willingness to follow all research procedures, including participation in all study visits and keeping a diary during the testing of preparations

Exclusion Criteria:

* Allergy to or suspicion of any ingredient in the test products
* menopause
* pregnancy, lactation
* in the past, surgery on the index finger / middle finger / ring finger of the right hand
* Disorders and deformities of the index finger, middle finger and ring finger of the right hand due to a malformation of the underlying bone, which would interfere with the evaluation of photographs or changes in the nails
* the presence of raised nails from the nail bed (onycholysis) on the index finger, middle finger and ring finger of the right hand
* supplementing the diet with dietary supplements containing CoQ10, biotin and other ingredients of the test product in the last three months before inclusion
* special eating habits used by a small part of the population (veganism, LCHF, calorie-restricted diets)
* diets prescribed by the medical profession
* uncontrolled metabolic and endocrine diseases
* Chronic dermatoses e.g. psoriasis, ichthyosis, various types of dermatitis, lichen planus, alopecia areata, scleroderma
* systemic diseases such as SLE, DLE, diabetes, neuropathy, peripheral artery disease
* have a known or suspected genetic condition that affects the nails (eg Darier's disease, nail patella syndrome, tuberculous sclerosis)
* the presence of anemia
* mental eating disorders
* mental incapacity that prevents proper understanding or cooperation
* sawing the surface of the nail plate or. polishing it in the last 6 months before inclusion and during the study
* any type of manicure involving gelling, artificial nails in the last 6 months before inclusion and during the study
* any type of classic manicure in the last month before inclusion and during the study
* change in the nail and hand care routine in the last month before inclusion and during the study
* change of dietary habits or dietary supplementation in the last 3 months before inclusion and during the study
* infections of the hands and nails on the hands (fungal, bacterial, viral)
* biting fingernails or cuticles
* mechanical irritation and damage to the nails,
* repeated prolonged exposure of the hands to water or repeated use of hand sanitizers,
* use of antimetabolites, retinoids, statins, antiretroviral drugs, fungicides in the last 3 months before inclusion and during the study
* changes in the use of hormonal preparations in the last 6 months before inclusion and during the study

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Change of frequency of nail fracture | 18 weeks
  Significant change of frequency of nail fracture from baseline in test group, in comparison to placebo group after 12 weeks of dietary supplementation with study product is expected. Frequency (number/day) of nail fracture will be assessed through diary of nail condition. For baseline nail fracture daily diary log will be kept for 4-6 weeks before dietary supplementation and for evaluation of treatment effects diary log will be kept from week 9 through 12 of the intervention.

SECONDARY OUTCOMES:
Change of the PGA score for assessment of the signs of brittle nails | 12 weeks
  Change of the signs of brittle nails from the initial state according to PGA score (physical global assessment score) after 12 weeks of supplementation with a test supplement compared to placebo. PGA scale of expression of changes on the nail: 0: no noticeable changes, 1: mild change, 2: mild / moderate change, 3: moderate change, 4: moderate / strong change, 5: strong change.
Change of the PGIA score for assessment of the signs of brittle nails | 12 weeks
  Change of the signs of brittle nails from the initial state according to PGIA score (physical global improvement assessment score) Improvement of brittle nail symptoms from baseline after 12 weeks of supplementation with a test supplement compared to a placebo product rated with a PGIA (physical global improvement assessment score): -1: worsening, 0: unchanged, 1: mild improvement, 2: moderate marked improvement, 3: strong improvement.
Change of the nail growth rate | 18 weeks
  Change in nail growth rate from baseline after 12 weeks of supplementation with a test supplement compared to placebo.
  For baseline nail growth rate nail will be market at week 0 and growth measured after 4-6 weeks, before start of the supplementation. For growth rate after supplementation nail will be market at week 8 and growth measured after 4 weeks of further supplementation.
Change in self-assessment of nail condition | 12 weeks
  Change in self-assessment of nail condition from baseline will be done at baseline and after 12 weeks of supplementation with a test supplement compared to a placebo product rated on a scale: 1 = very poor condition, 2 = poor condition, 3 = neither poor nor good condition, 4 = good condition, 5 = very good condition.
Change in expert assessment of nail condition | 12 weeks
  Change in expert assessment of nail condition from baseline will be done at baseline and after 12 weeks of supplementation with a test supplement compared to a placebo product rated on a scale: 1 = very poor condition, 2 = poor condition, 3 = neither poor nor good condition, 4 = good condition, 5 = very good condition.
Change of frequency in lamellar onychoschizia | 18 weeks
  Significant change of frequency of lamellar onychoschizia from baseline in test group, in comparison to placebo group after 12 weeks of dietary supplementation with study product is expected. Frequency of lamellar onychoschizia will be assessed through diary of nail condition. For baseline lamellar onychoschizia daily diary log will be kept for 4-6 weeks before dietary supplementation and for evaluation of treatment effects diary log will be kept from week 9 through 12 of the intervention.
Change of frequency of onychorrhexis | 18 weeks
  Significant change of frequency of onychorrhexis from baseline in test group, in comparison to placebo group after 12 weeks of dietary supplementation with study product is expected. Frequency of onychorrhexis will be assessed through diary of nail condition. For baseline onychorrhexis daily diary log will be kept for 4-6 weeks before dietary supplementation and for evaluation of treatment effects diary log will be kept from week 9 through 12 of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Katja Zmitek, PhD, Study Director — Visoka sola za storitve
Locations (1):
- Visoka sola za storitve, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No